CLINICAL TRIAL: NCT00323830
Title: Phase III Randomized Controlled Trial of Adjuvant Capecitabine/Cisplatin Chemotherapy and Chemoradiation Therapy for Gastric Adenocarcinoma
Brief Title: Phase III Randomized Trial of Adjuvant XP Chemotherapy and XP/RT for Resected Gastric Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-08-10
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Gastric Cancer; Surgery
Keywords: gastric cancer; radiotherapy; postoperative therapy; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; Radiotherapy

ARMS (2):
- capecitabine/cisplatin/radiotherapy (Experimental): postoperative XP/RT
  Interventions: Drug: Capecitabine, cisplatin, Radiotherapy (+/-)
- capecitabine/cisplatin (Active Comparator): postoperative XP
  Interventions: Drug: Capecitabine, cisplatin, Radiotherapy (+/-)

INTERVENTIONS:
Drug: Capecitabine, cisplatin, Radiotherapy (+/-) — Capecitabine, cisplatin + Radiotherapy (randomized)

SUMMARY:
The objective of the trial is to compare disease-free survival between adjuvant capecitabine/cisplatin alone vs capecitabine/cisplatin with radiotherapy (chemoradiation) in curatively resected gastric cancer patients.

DETAILED DESCRIPTION:
Although gastrectomy is the only potentially curative treatment in gastric cancer patients, the overall survival results remain unsatisfactory. The main factor accounting for high mortality rate is the relapse after surgical resection. During the past few decades, the principle of combined modality treatment has been developed and applied in practice for various solid tumors and gastric cancer has not been an exception. In an attempt to prevent recurrence and increase the cure rate of gastric cancer patients after surgery, multiple studies using variable modalities have been undertaken. One of the landmark study in adjuvant trials was the Intergroup study INT-0116, which reported a significant improvement in survival with the use of chemoradiation therapy after gastric resection of stage Ib to IV gastric cancers. Thereafter, the chemoradiation therapy has gained popularity and has been increasingly recognized as a standard of care in U.S. Nevertheless, the result from INT-0116 study has been challenged by the fact that the surgical treatment applied in the trial was gastrectomy with limited lymph node dissection (D0 or D1) in 90% of cases. Therefore, it is debatable whether adjuvant chemoradiation therapy can confer survival benefit in patients with extensive lymph node dissection.

It is still disputable if chemoradiotherapy after D2 can improve the results of D2 alone. Thus, the assessment of the effect of adjuvant chemoradiotherapy in D2 resected gastric cancer is essential.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven gastric adenocarcinoma
2. ≥ D2 resection
3. Stage IB(T1N1,T2bN0), II, IIIA, IIIB, IV(T4,N3 포함, M1 lymph node 제외)
4. 18 ≤ age ≤ 75
5. ECOG 0-2
6. No distant metastasis
7. Adequate bone marrow functions (ANC ≥ 1,500/ul, blood platelet ≥ 100,000/ul, haemoglobin ≥ 10g/dl)
8. Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
9. liver functions (serum bilirubin ≤ 1.5mg/dl, AST/ALT ≤ 3 times(normal value)
10. Written informed consent

Exclusion Criteria:

1. Previous history of immunotherapy, chemotherapy, radiotherapy for gastric cancer
2. Active infection requiring antibiotics
3. Pregnant, lactating women
4. Psychiatric illness, epileptic disorders
5. Concurrent systemic illness not appropriate for chemotherapy
6. Resection margin (+)
7. Pathologic stage IA
8. History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma
9. M1 lymph node (+)
10. D0, D1 resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
disease free survival | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park SH, Sohn TS, Lee J, Lim DH, Hong ME, Kim KM, Sohn I, Jung SH, Choi MG, Lee JH, Bae JM, Kim S, Kim ST, Park JO, Park YS, Lim HY, Kang WK. Phase III Trial to Compare Adjuvant Chemotherapy With Capecitabine and Cisplatin Versus Concurrent Chemoradiotherapy in Gastric Cancer: Final Report of the Adjuvant Chemoradiotherapy in Stomach Tumors Trial, Including Survival and Subset Analyses. J Clin Oncol. 2015 Oct 1;33(28):3130-6. doi: 10.1200/JCO.2014.58.3930. Epub 2015 Jan 5. PMID 25559811